CLINICAL TRIAL: NCT06636773
Title: Effectiveness of the Addition of Yoga to a Behavioral Weight Loss Intervention for Adults With Overweight or Obesity (MOVE for Health)
Brief Title: Comparision of Aerobic Exercise to Aerobic Plus Yoga Exercise for Weight Loss in Adults With Overweight or Obesity.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, John M. Jakicic, PhD, Professor, University of Kansas Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00160080; R01DK135735-01A1 (NIH)
Record Dates: First submitted 2024-10-04; First posted 2024-10-15 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Obesity and Overweight
Keywords: obesity; overweight; exercise; physical activity; yoga; weight loss
MeSH Terms: conditions — Obesity; Overweight; Motor Activity; Weight Loss | interventions — Diet; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral Weight Loss Plus Aerobic Physical Activity (Experimental): The intervention is a 12-month behavioral intervention focused on modifying eating behaviors and physical activity. Participants will be provided weekly group-based behavioral session for months 1-6, with these sessions being offered twice per month during months 7-12. Participants will be instructed to self-monitor their weight, eating behaviors, and physical activity. A reduced energy diet ranging from 1200-2100 kilocalories per day will be recommended for participants. Physical activity will be recommended in the form of aerobic types of activity such as brisk walking and will progress from an initial amount of 100 minutes per week to 300 minutes per week across the initial 6 months of the intervention, with this level of physical activity continuing to be recommended between months 7-12.
  Interventions: Behavioral: Diet; Behavioral: Aerobic Exercise; Behavioral: Behavioral Sessions
- Behavioral Weight Loss Plus Aerobic Physical Activity and Yoga (Experimental): The intervention is a 12-month behavioral intervention focused on modifying eating behaviors and physical activity. Participants will be provided weekly group-based behavioral session for months 1-6, with these sessions being offered twice per month during months 7-12. Participants will be instructed to self-monitor their weight, eating behaviors, and physical activity. A reduced energy diet ranging from 1200-2100 kilocalories per day will be recommended for participants. Physical activity will be recommended in the form of aerobic types of activity such as brisk walking combined with yoga. Aerobic activity will progress from an initial amount of 60 minutes per week to 180 minutes per week across the initial 6 months of the intervention, with this level continuing to be recommended between months 7-12. Yoga will progress from 40 minutes per week to 120 minutes per week across the initial 6 months of the intervention, with this level continuing to be recommended between months 7-12.
  Interventions: Behavioral: Diet; Behavioral: Behavioral Sessions; Behavioral: Aerobic + Yoga Exercise

INTERVENTIONS:
Behavioral: Diet — A reduced energy diet ranging from 1200-2100 kilocalories per day will be recommended for participants.
Behavioral: Aerobic Exercise — Physical activity will be recommended in the form of aerobic types of activity such as brisk walking and will progress from an initial amount of 100 minutes per week to 300 minutes per week across the initial 6 months of the intervention, with this level of physical activity continuing to be recommended between months 7-12.
  Arms: Behavioral Weight Loss Plus Aerobic Physical Activity
Behavioral: Behavioral Sessions — Participants will be provided weekly group-based behavioral session for months 1-6, with these sessions being offered twice per month during months 7-12 to assist in supporting recommended changes in energy intake (diet) and physical activity.
Behavioral: Aerobic + Yoga Exercise — Physical activity will be recommended in the form of a combination of aerobic types of activity, such as brisk walking, and yoga. Aerobic activity will progress from 60 minutes per week to 180 minutes per week across the initial 6 months of the intervention. Yoga will progress from 40 minutes per week to 120 minutes per week across the initial 6 months of the intervention. When combined this will progress from a total of 100 minutes per week to 300 minutes per week across the initial 6 months of treatment. This level of physical activity will continue to be recommended between months 7-12.
  Arms: Behavioral Weight Loss Plus Aerobic Physical Activity and Yoga

SUMMARY:
The goal of this clinical trial is to learn whether adding yoga exercise to a behavioral weight loss intervention improves weight loss in adults with overweight or obesity. It will also provide information about whether this approach to weight loss has additional benefits on other health and fitness measurements. The main questions it aims to answer are:

* Is there a difference in weight loss between the behavioral program that includes aerobic exercise plus yoga compared to the behavioral program that includes only aerobic exercise?
* Is there a difference in how much physical activity is completed between the behavioral program that includes aerobic exercise plus yoga compared to the behavioral program that includes only aerobic exercise?
* Is there a difference in the change in body composition (fat mass, lean body mass) between the behavioral program that includes aerobic exercise plus yoga compared to the behavioral program that includes only aerobic exercise?
* Is there a difference in the change in cardiorespiratory fitness the behavioral program that includes aerobic exercise plus yoga compared to the behavioral program that includes only aerobic exercise?
* Is there a difference in the change in muscle strength between the behavioral program that includes aerobic exercise plus yoga compared to the behavioral program that includes only aerobic exercise?
* Is there a difference in the change in resting blood pressure between the behavioral program that includes aerobic exercise plus yoga compared to the behavioral program that includes only aerobic exercise?
* Is there a difference in the change in food intake or eating behaviors between the behavioral program that includes aerobic exercise plus yoga compared to the behavioral program that includes only aerobic exercise?
* Is there a difference in the change in feelings of stress or mood between the behavioral program that includes aerobic exercise plus yoga compared to the behavioral program that includes only aerobic exercise?
* Is there a difference in the change in sleep between the behavioral program that includes aerobic exercise plus yoga compared to the behavioral program that includes only aerobic exercise?
* Is there a difference in the change in mindfulness between the behavioral program that includes aerobic exercise plus yoga compared to the behavioral program that includes only aerobic exercise?

Participants will:

* Participate in a weight loss program for a period of 12 months that involves attending behavioral weight loss sessions. This involves coming to a session at the research center weekly for the initial 6 months and then every other week for the remaining 6 months.
* Attempt to reduce the amount of food that they eat to reduce the calories they consume.
* Participate in a combination of aerobic exercise plus yoga or just aerobic exercise.
* Keep a record of the food they consume, use a digital scale provided to them, and wear an activity tracker provided to them for the period of 12 months.
* Visit the clinical before starting the weight loss program, after 3 months, 6 months, 9 months, and 12 months to complete measurements of their weight and other measurements to monitor their progress.
* Complete exercise sessions in the clinic between weeks 2-6, at month 6, and at month 12 to provide information about how they response to a single session of exercise.

ELIGIBILITY:
Inclusion Criteria:

* Both males and females of all race/ethnic groups are eligible for participation in this study.
* at least 18 years of age. The investigators will not limit enrollment based on an upper age provided that the participant meets the other eligibility requirements.
* Body mass index (BMI) of at least 25.0 kg/m2. The investigators will not limit enrollment based on an upper BMI level provided that the participant meets the other eligibility requirements. However, maximal weight to be eligible will be 350 pounds to meet the weight requirements for the equipment that will be used in this study.
* Ability to provide informed consent prior to participation in this study.
* Ability to provide clearance from their primary care physician to engage in the diet and physical activity components of the weight loss intervention.

Exclusion Criteria:

* Report moderate-to-vigorous exercise on >3 days/week or a total of >60 min/week over the past 3 months.
* Engaging in any style of yoga on an average of at least 1 day/week over the past 3 months.
* Report weight loss of 3% or more or participating in a weight reduction diet in the past 3 months.
* Currently prescribed an anti-obesity medication.
* Females who are pregnant or breastfeeding or reporting a planned pregnancy during the study period.
* History of bariatric surgery.
* Report a current medical condition or treatment for a medical condition that could affect body weight.
* Current congestive heart failure, angina, uncontrolled arrhythmia, symptoms indicative of an increased acute risk for a cardiovascular event, prior myocardial infarction, coronary artery bypass grafting or angioplasty, conditions requiring chronic anticoagulation (i.e., recent or recurrent DVT).
* Resting systolic blood pressure of 160 mmHg or more or resting diastolic blood pressure of 100 mmHg or more. If medicated for blood pressure control, the medication dose needs to be stable for at least 6 months.
* Eating disorders that would contraindicate weight loss or physical activity.
* Alcohol or substance abuse.
* Current psychological condition that is untreated, hospitalization for a psychological condition within the past 12 months, or not being on a stable dose of treatment for at least 6 months.
* Report plans to relocate to a location not accessible to the study site or having employment, personal, or travel commitments that prohibit attendance at scheduled intervention sessions or assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Estimated)
Dates: Start 2025-01-03 (Actual); Primary Completion 2028-11-30 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
Body Weight | 0, 3, 6, 9, 12 months
  Body weight will be assessed in duplicate using a calibrated digital scale to the nearest 0.1 kg.

SECONDARY OUTCOMES:
Body Mass Index | 0, 3, 6, 9, 12 months
  Measurements of weight and height will be used to compute BMI (kg/m2).
Percent body fat | 0, 6, 12 months
  Percent body fat will be assessed using a total body scan from dual-energy x-ray absorptiometry (DXA).
Body Fat Mass | 0, 6, 12 months
  Body fat mass (kg) will be assessed using a total body scan from dual-energy x-ray absorptiometry (DXA).
Lean Body Mass | 0, 6, 12 months
  Lean body mass (kg) will be assessed using a total body scan from dual-energy x-ray absorptiometry (DXA).
Bone mineral content | 0, 6, 12 months
  Bone mineral content (grams) will be assessed using a total body scan from dual-energy x-ray absorptiometry (DXA).
Waist Circumference | 0, 6, 12 months
  Circumference measures of the waist taken horizontally at both the iliac crest and the umbilicus will be performed.
Cardiorespiratory Fitness | 0, 6, 12 months
  Cardiorespiratory fitness will be represented as milliliters of oxygen consumed per kilogram of body weight per minute (ml/kg/min) measured with a metabolic cart during a submaximal graded exercise test that is terminated when the participant achieves 85% of age-predicted maximal heart rate.
Cardiorespiratory Fitness | 0, 6, 12 months
  Cardiorespiratory fitness will be represented as total liters of oxygen consumed per minute (L/min) measured with a metabolic cart during a submaximal graded exercise test that is terminated when the participant achieves 85% of age-predicted maximal heart rate.
Cardiorespiratory Fitness | 0, 6, 12 months
  Cardiorespiratory fitness will be the duration measured in minutes to achieve 85% of age-predicted maximal heart rate during a submaximal graded exercise test performed on a treadmill.
Energy Intake (Dietary Intake) | 0, 3, 6, 9, 12 months
  Energy Intake (Dietary Intake) expressed as kilocalories eaten per day (kcal/day) will be measured using the Diet History Questionnaire (DHQ) developed by NCI. A higher score represents more calories eaten.
Dietary Cognitive Restraint | 0, 3, 6, 9, 12 months
  Dietary cognitive restraint will be measured using from 21 items on the 3-Factor Eating Questionnaire. The range of possible scores is 0 to 20, with a higher score representing high dietary cognitive restraint.
Dietary Disinhibition | 0, 3, 6, 9, 12 months
  Dietary disinhibition will be measured using from 16 items on the 3-Factor Eating Questionnaire. The range of possible scores is 0 to 16, with a higher score representing high dietary disinhibition.
Hunger | 0, 3, 6, 9, 12 months
  Hunger will be measured using from 15 items on the 3-Factor Eating Questionnaire. The range of possible scores is 0 to 15, with a higher score representing high hunger.
Weight Loss Strategies | 0, 3, 6, 9, 12 months
  Weight Loss Strategies will be measured using the Weight Control Strategies Scale that includes 30 items. A higher score represents engaging in more weight control strategies.
Weight Loss Strategies | 0, 3, 6, 9, 12 months
  Weight Loss Strategies will be measured using the Eating Behavior Inventory that includes 26 items with each measured on a 5-point scale. A higher score represents engaging in more weight loss strategies.
Mood/Affect | 0, 3, 6, 9, 12 months
  The Positive and Negative Affect Schedule (PANAS) will be used to assess mood/affect which includes 20 items measured on a 5-point scale. A higher score represents a higher degree of either positive or negative affect.
Perceived Stress | 0, 3, 6, 9, 12 months
  Perceived Stress Scale (PSS) will assess a global appraisal of perceived stress, which includes 10 items each score on a 5-point scale. A higher score represents higher perceived stress.
Depressive Symptoms | 0, 3, 6, 9, 12 months
  Centers for Epidemiological Studies Depression Scale (CES-D) will assess depressive symptoms. This includes 10 items scored on a scale of 0-4, with a higher score representing higher depressive symptoms.
Mindfulness | 0, 3, 6, 9, 12 months
  The Mindful Attention Awareness Scale is used to measure mindfulness. It contains 15 items scored on a 1-6 scale, and a higher score represents more mindfulness.
Mindfulness Practice | 0, 3, 6, 9, 12 months
  The Five-Facet Mindfulness Questionnaire will be used to assess mindfulness and mindfulness practice. It contains 39 items scored on a 5-point scale, and a higher score represents more mindfulness practice.
Sleep | 0, 3, 6, 9, 12 months
  Sleep will be assessed using the Pittsburgh Sleep Quality Index. The sum of 7 domains, each scored on a 0-3 scales, provide a total score that ranges from 0-21. A higher score indicates greater sleep disturbance.
Acute Physical Activity Test - perceived distress | Between weeks 2-6, at 6 months, at 12 months
  Perceived distress will be measured using a questionnaire that includes 12 items scored on a 7-point scale.
Acute Physical Activity Test - Mood | Between weeks 2-6, at 6 months, at 12 months
  Mood will be measured using a questionnaire. The Positive and Negative Affect Schedule (PANAS) will be used to assess mood/affect which includes 20 items measured on a 5-point scale. A higher score represents a higher degree of either positive or negative affect.
Acute Physical Activity Test - Sleepiness | Between weeks 2-6, at 6 months, at 12 months
  Sleepiness will be measured using on a 9-point scale with a higher score representing more sleepiness.
Acute Physical Activity Test - Hunger | Between weeks 2-6, at 6 months, at 12 months
  Hunger will be measured using a 100 mm visual analog scale, with a higher score representing more hunger.
Acute Physical Activity Test - Cortisol | Between weeks 2-6, at 6 months, at 12 months
  Cortisol will be measured from a blood sample using a commercially available assay.

OTHER OUTCOMES:
Medication History | 0, 3, 6, 9, 12 months
  A questionnaire developed specifically for this study will be used to assessment medication history. The data collected include the type of medication, dose of medication, and frequency that the medication is taken, and what condition the medication is indicated to treat.
Lifestyle and Health History | 0 months (prior to randomization)
  A questionnaire developed specifically for this study that is conducted as an interview will be used to assess lifestyle and health factors to describe the sample for this study. The score is either "yes" or "no" identifying the presences of a lifestyle or health factor.
Adverse and Serious Adverse Events | 0, 3, 6, 9, 12 months and at other times when reported by the participant
  Participants will be queried using a survey developed specifically for this study will be used to assess for adverse events and serious adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: John M. Jakicic, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: Yes
The summary data for each of the study outcomes and other additional demographic characteristics will be made available. The Study Protocol (which includes the statistical analysis plan), Manual of Procedures, Data Collection Forms, and a Data Dictionary to explain the data variables will be provided.
Supporting Information: Study Protocol, SAP
Time Frame: The data will be made available no later than the time of an associated publication of study outcomes or at the end of the performance period, whichever comes first. The data provided to the repository will be available indefinitely while that repository continues to exist.
Access Criteria: The information included with the IPD will be made available to appropriate individuals only after the requester confirms their willingness to comply with an appropriate "Data Use Agreement" that complies with NIH policies, the policies of the institution where the study has been conducted, and the elements of informed consent.